CLINICAL TRIAL: NCT06297889
Title: Effects of Core Strength Training on Physical Fitness and Field Hockey Skills Performance Among Youth Male Field Hockey Players in Gansu, China
Brief Title: Effect of Core Strength Training on the Physical Fitness and Skills of Youth Field Hockey Players in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, MA HUCHENG, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: Ma Hucheng
Record Dates: First submitted 2024-02-19; First posted 2024-03-07 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Player
Keywords: Core Strength Training; Physical Fitness; skills performance

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group engaged in the core strength training segment of the intervention specifically devised for this study, whereas the control group underwent conventional strength training activities.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core strength training interventions for 1-6 weeks (Experimental): Core strength training: Experiment: Experimental Group: Core Strength Training for 1-6 Weeks.Participants undergo a one-hour training session three times a week for 1- 6 weeks, incorporating a 15-minute warm-up followed by 45 minutes of targeted core strength training.
  Interventions: Behavioral: core strength training 1-6weeks; Behavioral: core strength training 7-12weeks
- Core strength training interventions for 7-12 weeks (Experimental): Core strength training: Experiment: Experimental Group: Core Strength Training for 7-12 Weeks.Participants undergo a one-hour training session three times a week for 7-12 weeks, incorporating a 10-minute warm-up followed by 50 minutes of targeted core strength training.
  Interventions: Behavioral: core strength training 1-6weeks; Behavioral: core strength training 7-12weeks

INTERVENTIONS:
Behavioral: core strength training 1-6weeks — Behaviour: core strength training intervention for 1-6 weeks. Experimental: The experimental group performed core strength training during weeks 1-3. Subjects were first provided with basic information, familiarised with the content of the first phase of core strength training and watched a core strength video to understand its importance. The initial intervention was designed to ensure that subjects were proficient in core strength training, including warm-up and stretching patterns. During weeks 4-6, subjects will be supervised and assisted and a test will be organised at the end of week 6. Variables related to physical fitness and skills were recorded to assess whether core strength training improved physical fitness and skills.
Behavioral: core strength training 7-12weeks — Behaviour: core strength training intervention #7-12 weeks#.
  Experimental: Weeks 7-9 were the experimental group:
  Continued to warm up before each training session. The training content will increase in difficulty during this phase, and the supervisor should explain the training content and watch videos of the movements prior to training and prepare the training equipment in advance to protect the athlete from injury. Weeks 10-12: This is an advanced stage, requiring equipment and difficult movements to complete, please supervisors to arrange personnel to do a good job of protection to ensure that the subjects can complete the training tasks. A test will be conducted the day after Week 12 to measure the athlete's physical fitness and skills.

SUMMARY:
Hockey, tracing its origins back to 2000 BC, has undergone substantial evolutionary transformations throughout the centuries. Initially known by various names, the game transitioned to its modern form approximately 50 years ago, when matches were conducted on grass fields with wooden sticks. In contemporary international hockey, there has been a notable shift towards artificial grass, cultivating a dynamic and fast-paced game that places heightened demands on individual skills, tactical acumen, and physical fitness. This evolution reflects a continuous adaptation, seamlessly blending tradition with cutting-edge equipment and hybrid playing grounds.

Against this backdrop, modern-day hockey programs have metamorphosed into rigorous and demanding training regimes. Athletes engaged in these programs are required not only to demonstrate outstanding physical fitness but also exhibit a high level of proficiency in the nuanced skills essential for competitive play. As hockey continues its progressive trajectory, athletes partaking in these programs must meet elevated standards, underscoring the imperative integration of both exceptional fitness levels and precise skill execution.

Despite the growing emphasis on the physical and skill dimensions of hockey, a literature review uncovered a dearth of research specifically focusing on core strength training for hockey players. While core strength training has demonstrated efficacy in improving physical fitness and skill performance among athletes in other team sports, its applicability to hockey players remains underexplored. Moreover, no studies have systematically examined the impact of core strength training on the two critical variables of physical fitness and skill performance in hockey players.

To address this research gap, the present study sought to investigate the effects of core strength training on the physical fitness and skill performance of youth hockey players in Gansu Province, China. By doing so, this study not only contributes valuable insights to the existing body of literature but also furnishes theoretical support for the development of hockey sport programs. The findings are anticipated to inform targeted interventions aimed at enhancing athletes' physical fitness and skill performance, ultimately fostering the progression of hockey programs within the sporting landscape of China.

DETAILED DESCRIPTION:
present study employed a two-group design consisting of a Control Group (CG) and an Experimental Group (EG). The training trial extended over 12 weeks, with sessions scheduled three (3) times weekly, each lasting one hour (1). The training regimen was organized into four distinct stages：beginner (1-3 weeks), intermediate (4-6 weeks), upper intermediate (7-9 weeks) and advanced (10-12 weeks).

Since the participants were young male athletes instead of adults, special attention was devoted to calibrating training intensity. Consistent with existing research, the intensity of strength training was designed to gradually escalate from low to high, adhering to the principle of training specificity (Faigenbaum et al., 2012; Harries et al., 2016). The recommended intensity levels were set at 60% of the one-repetition maximum (1RM), progressing to 70% and 80% 1RM(Brown,2007). This careful structuring of the program aimed to adapt the core strength training to the physiological characteristics and needs of youth athletes, ensuring both efficacy and safety throughout the trial period.Therefore, I invite experts to evaluate and score the experiment design, helping me do this experiment better.

ELIGIBILITY:
Inclusion Criteria:

-

This study was conducted with male hockey players from Gansu Sports School and Linxia Sports School. Before recruiting the subjects, the researcher needed to inform the subjects of the proposed study and what they needed to participate in. After informing the subjects, the subjects will be allowed to ask questions. Various criteria and requirements for participation in this study are explained during the session. The inclusion criteria for potential participants were as follows:

1. Male
2. Aged 15 to 17 years
3. Reside in Gansu Province, China
4. Healthy
5. Two years of training experience

Exclusion Criteria:

1. on medication which may affect body composition and muscles activity like Diabetes Mellitus
2. Currently participating in regular resistance training

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Power test | pretest, week 6, week 12
  1.Power: Athletes perform the standing medicine ball throw test by turning their body to one side, bending their knees slightly, and forcefully throwing a 2 (kg) medicine ball forward. The test measures the vertical distance between the point of impact of the ball and the marking line. The athlete performs three trials on each side and the performance is measured in (m), e.g., (10.78 m on the left side) the best performance is recorded to assess functional power.
Speed test | pretest, week 6, week 12
  2.Speed: The athlete performs 25 (m) and 50 (m) sprints from the bottom line of the hockey rink using Speed Smart infrared speed measuring equipment placed at a specified distance. The athlete stands 0.1 (m) from the device and sprints forward as hard as he/she can, with the infrared timing system automatically recording the time it takes the athlete to complete the 25 (m) and 50 (m) distances. Each athlete performs three trials and the performance is based on (m/s). The shorter the time, the better the acceleration and speed.

CONTACTS AND LOCATIONS:
Overall Officials: Hucheng Ma, PHD, Principal Investigator — University Putra Malaysia
Locations (1):
- Ma Hucheng, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Result] Axel TA, Crussemeyer JA, Dean K, Young DE. Field Test Performance of Junior Competitive Surf Athletes following a Core Strength Training Program. Int J Exerc Sci. 2018 Jun 1;11(6):696-707. doi: 10.70252/XHXE2254. eCollection 2018. PMID 29997737
- [Result] Faigenbaum AD, McFarland JE, Herman RE, Naclerio F, Ratamess NA, Kang J, Myer GD. Reliability of the one-repetition-maximum power clean test in adolescent athletes. J Strength Cond Res. 2012 Feb;26(2):432-7. doi: 10.1519/JSC.0b013e318220db2c. PMID 22233786
- [Result] Willardson, J. M. (2013). Developing the core. Human Kinetics.
- See also: Sources of training programmes — http://books.google.com.my/books?hl=zh-CN&lr=&id=MvB6DwAAQBAJ&oi=fnd&pg=PR7&dq=Willardson,+J.+M.+(2013).%C2%A0Developing+the+core.+Human+Kinetics.&ots=UO-TaVWJkq&sig=JvjEmYfHZAWciv1GIi0DAw_uUCs&redir_esc=y#v=onepage&q=Willardson%2C%20J.%20M.%20(2013).%C2%A0Developing%20the%20core.%20Human%20Kinetics.&f=false